CLINICAL TRIAL: NCT05399732
Title: A Randomized, Case Controlled Clinical Trial Evaluating the Efficiency and Safety of Luspatercept Plus Cyclosporine Versus Cyclosporine in Newly Diagnosed Transfusion Independent Non-severe Aplastic Anemia (NSAA).
Brief Title: Efficacy and Safety in Transfusion Independent Non-severe Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bing Han (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Bing Han, professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HanB-NSAA-lus
Record Dates: First submitted 2022-05-24; First posted 2022-06-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Aplastic Anemia
Keywords: NSAA; luspatercept; ORR; non-transfusion dependent
MeSH Terms: conditions — Anemia, Aplastic | interventions — luspatercept; Cyclosporine

STUDY DESIGN:
Intervention Model Description: Cyclosporine soft capsules（25mg） are produced by North China pharmaceutical Group Corporation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- efficiency and safety in luspatercept plus cyclosporine (Experimental): luspatercept is at a dose of 1.0 mg per kilogram of body weight, administered subcutaneously every 3 weeks，and cyclosporine is at a dose of 3~5mg/kg /day for at least 6 months.
  Interventions: Drug: Luspatercept; Drug: Cyclosporine
- controll group in cyclosporine alone (Active Comparator): cyclosporine is at a dose of 3~5mg/kg /day for at least 6 months.
  Interventions: Drug: Cyclosporine

INTERVENTIONS:
Drug: Luspatercept — Patients in each group will be treated for at least 6 months and continue the treatment for an additional 6 months unless disease progress or have intolerable side effects.
  Arms: efficiency and safety in luspatercept plus cyclosporine
Drug: Cyclosporine — Cyclosporine was administered at a 3-5 mg/(kd/d) and maintained at a 100-200 ng/ml trough plasma concentration.
  Other Names: Ciclosporin; Cyclosporin

SUMMARY:
Aplastic anemia (AA) is a rare bone marrow failure disease characterized by bone marrow hypocellularity and peripheral blood pancytopenia. AA is divided into severe AA (SAA) and non-severe AA (NSAA) based on the degree of cytopenia. The first line therapy for SAA or transfusion dependent NSAA is either immunosuppression therapy (IST) or hematopoietic stem cell transplantation (HSCT). Little attention has been paid to patients with anemia but not transfusion dependent, whose quality of life is significantly impaired due to the anemia and other complications.

DETAILED DESCRIPTION:
Recombined human erythropoietin (rhEPO) has been shown to increase the erythroid response and response rate when combined with IST for patients with newly diagnosed AA, either SAA or NSAA. Different from rhEPO, luspatercept is a recombinant fusion protein that binds to select transforming growth factor β superfamily ligands and enhances late-stage erythropoiesis, and has been shown the promising efficiency in the erythropoiesis in patients with lower risk myelodysplastic syndrome (MDS) in the phase II and III clinical trials. This randomized control study aimed to compare the 6-month efficacy and safety of the combination of luspatercept and cyclosporine versus cyclosporine monotherapy in patients with newly diagnosed transfusion independent NSAA.

ELIGIBILITY:
Inclusion Criteria:

1. age≥18 year-old;
2. hemoglobin level between 60g/L~10 g/dL;
3. newly diagnosed patients have at least one of the followings: #absolute neutrophil count <1.5×109/L, #platelet count < 30×109/L, # hemoglobin level < 100g/L;
4. with normal baseline liver and kidney function;
5. with no active infection; are not pregnant or nursing;
6. agree to sign consent forms;
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Exclusion Criteria:

1. Congenital aplastic anemia;
2. Presence of chromosomal aberration;
3. Evidence of a clonal hematologic bone marrow disorder (MDS, AML) on cytogenetics;
4. Presence with PNH clone ≥50%;
5. Patients received HSCT before;
6. Uncontrolled infection or bleeding with standard treatment;
7. Allergic to luspatercept CsA or accessories;
8. HIV, HCV or HBV active infection or liver cirrhosis or portal hypertension;
9. Patient with QTcF (Fridericia's QT correction formula) at screening <450 msec, or<480 msec with bundle branch block, as determined via the mean of a triplicate ECG and assessed at site, unstable angina pectoris, uncontrolled hypertension(>180/100mmHg)#pulmonary artery hypertension;
10. Have any concomitant malignancies within 5 years expect for local basal cell carcinoma of the skin;
11. Past history of thromboembolic event, heart attack or stroke (including anti-phospholipid antibody syndrome) and current use of anticoagulants;
12. Pregnant or nursing (lactating) woman;
13. Have attended other clinical trials within 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
overall response rate (ORR) | 6 month
  Overall Response Rate (ORR) Defined as the Number of Participants Who Met the Criteria of Either Complete Response (CR) or Partial Response (PR); HR defined as a hemoglobin increase from baseline of ≥1.5 g/dL for ≥2 weeks (in the absence of RBC transfusions)

SECONDARY OUTCOMES:
Hematologic response-erythroid（HR-E) | 6 month
  HR is defined as a hemoglobin increase from baseline of ≥1.5 g/dL for ≥2 weeks (in the absence of RBC transfusions
side effects | 1 year
  Safety analyses include assessments of the incidence and severity of adverse events; all adverse events that occurred or worsened during the treatment period will be reported, as well as adverse events that occurred later but are considered by the investigator to be related to the trial drug.
predictive factors | 6 month
  Predictors analyses will evaluate the relationship between the effect of these two treatments with molecular mutations PIGA and BCOR and BCORL1 and EPO level.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data would be accepted upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 10years
Access Criteria: email request

REFERENCES:
- [Background] Howard SC, Naidu PE, Hu XJ, Jeng MR, Rodriguez-Galindo C, Rieman MD, Wang WC. Natural history of moderate aplastic anemia in children. Pediatr Blood Cancer. 2004 Oct;43(5):545-51. doi: 10.1002/pbc.20131. PMID 15382271
- [Background] Zhang ML, Chen WS, Han B. [Evaluation of the efficacy of cyclosporin A combined with recombined human thrombopoietin for treating patients with non-severe aplastic anemia]. Zhonghua Xue Ye Xue Za Zhi. 2020 Aug 14;41(8):637-642. doi: 10.3760/cma.j.issn.0253-2727.2020.08.004. Chinese. PMID 32942816
- [Background] Chen WS, Zhang ML, Han B. [Evaluation of the Efficacy of Cyclosporin A Combined with Recombined Human Erythropoietin in the Treatment of Patients with Chronic Aplastic Anemia]. Zhongguo Yi Xue Ke Xue Yuan Xue Bao. 2021 Oct;43(5):736-742. doi: 10.3881/j.issn.1000-503X.13201. Chinese. PMID 34728034
- [Background] Furlong E, Carter T. Aplastic anaemia: Current concepts in diagnosis and management. J Paediatr Child Health. 2020 Jul;56(7):1023-1028. doi: 10.1111/jpc.14996. Epub 2020 Jul 3. PMID 32619069
- [Background] Desmond R, Townsley DM, Dunbar C, Young NS. Eltrombopag in aplastic anemia. Semin Hematol. 2015 Jan;52(1):31-7. doi: 10.1053/j.seminhematol.2014.10.002. Epub 2014 Oct 31. PMID 25578417
- [Background] Matsuda K, Koya J, Arai S, Nakazaki K, Nakamura F, Kurokawa M. Cyclosporine Therapy in Patients with Transfusion-independent Non-severe Aplastic Anemia: A Retrospective Analysis. Intern Med. 2019 Feb 1;58(3):355-360. doi: 10.2169/internalmedicine.1372-18. Epub 2018 Aug 24. PMID 30146592
- [Background] Drexler B, Passweg J. Current evidence and the emerging role of eltrombopag in severe aplastic anemia. Ther Adv Hematol. 2021 Mar 3;12:2040620721998126. doi: 10.1177/2040620721998126. eCollection 2021. PMID 33747425